CLINICAL TRIAL: NCT00851890
Title: A Blinded, Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Multiple Doses of ABT-333 Alone and in Combination With Pegylated Interferon (pegIFN) and Ribavirin (RBV) in Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Multiple Doses of ABT-333 Alone and in Combination With Pegylated Interferon (pegIFN) and Ribavirin (RBV) in Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-380
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2014-12

CONDITIONS: Chronic Hepatitis C Virus Infection
MeSH Terms: interventions — dasabuvir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ABT-333 (300 mg) twice daily (BID) + pegIFN/RBV (Experimental): Hepatitis C virus (HCV) positive, treatment-naive participants received 300 mg ABT-333 BID for 2 days followed by 300 mg ABT-333 BID with pegylated interferon/ribavirin (pegIFN/RBV) for 26 days. Pegylated interferon was administered at 180 μg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-333; Drug: Pegylated interferon; Drug: Ribavirin
- ABT-333 (600 mg) twice daily (BID) + pegIFN/RBV (Experimental): Hepatitis C virus (HCV) positive, treatment-naive participants received 600 mg ABT-333 BID for 2 days followed by 600 mg ABT-333 BID with pegylated interferon/ribavirin (pegIFN/RBV) for 26 days. Pegylated interferon was administered at 180 μg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-333; Drug: Pegylated interferon; Drug: Ribavirin
- ABT-333 (1200 mg) once daily (QD) + pegIFN/RBV (Experimental): Hepatitis C virus (HCV) positive, treatment-naive participants received 1200 mg ABT-333 QD for 2 days followed by 1200 mg ABT-333 QD with pegylated interferon/ribavirin (pegIFN/RBV) for 26 days. Pegylated interferon was administered at 180 μg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-333; Drug: Pegylated interferon; Drug: Ribavirin
- Placebo + pegIFN/RBV (Placebo Comparator): Hepatitis C virus (HCV) positive, treatment-naïve participants received matching placebo once daily (QD) or twice daily (BID) for 2 days followed by placebo QD or BID with pegylated interferon/ribavirin (pegIFN/RBV) for 26 days. Pegylated interferon was administered at 180 μg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Other: Placebo for ABT-333; Drug: Pegylated interferon; Drug: Ribavirin

INTERVENTIONS:
Drug: ABT-333 — 50 mg capsules
  Other Names: dasabuvir
  Arms: ABT-333 (1200 mg) once daily (QD) + pegIFN/RBV; ABT-333 (300 mg) twice daily (BID) + pegIFN/RBV; ABT-333 (600 mg) twice daily (BID) + pegIFN/RBV
Other: Placebo for ABT-333 — Capsule
  Arms: Placebo + pegIFN/RBV
Drug: Pegylated interferon — Syringe, 180 µg/0.5 mL for subcutaneous injections administered weekly
Drug: Ribavirin — 200 mg tablet dosed at 1000 or 1200 mg daily divided twice a day

SUMMARY:
The purpose of this study was to assess the safety, tolerability, pharmacokinetics and antiviral activity of ABT-333 (also known as dasabuvir) in treatment-naïve, hepatitis C virus (HCV)-infected participants.

DETAILED DESCRIPTION:
This was a Phase 2a, blinded, randomized, placebo-controlled clinical trial in hepatitis C virus (HCV)-infected adults with 2 planned sequential evaluations, Part 1 and Part 2. The study evaluated the safety, tolerability, antiviral activity, and pharmacokinetics of ABT-333 or placebo monotherapy, followed by 26 days of ABT-333 or placebo with pegylated interferon a-2a (pegIFN) and ribavirin (RBV) combination therapy. Review of safety and efficacy in Part 1 of the study showed similar response rates across ABT-333 doses so Part 2 of the study was not performed. The study also assessed emergence of resistant HCV in conjunction with kinetics of viral load decay and rebound in treatment-naïve, HCV-infected participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided written consent.
* If female, participant is postmenopausal or surgically sterile.
* If male, must be practicing two effective methods of birth control.
* Participant is hepatitis C virus (HCV) genotype 1 with HCV ribonucleic acid levels >50,000 IU/mL.
* Participants must demonstrate chronic hepatitis C infection for at least 6 months prior to study enrollment.
* Participants must have a liver biopsy with histology consistent with HCV-induced liver damage, and with no evidence of cirrhosis or liver pathology due to any cause other than chronic HCV.
* Condition of general good health other then HCV infection.
* Participants with a history of thyroid disease must have a thyroid stimulating hormone (TSH) value in the normal range.

Exclusion Criteria:

* No prior history of receiving therapy for HCV infection.
* Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus antibody (HIV Ab).
* Pregnant or breastfeeding females or male partners of women who are pregnant.
* History of seizures or cancer.
* History of major depressive disorder within 2 years.
* Any current or past history of cirrhosis.
* Any cause of liver disease other than chronic HCV infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MD, Study Director — AbbVie
Locations (8):
- United States (7):
  - Site Reference ID/Investigator# 16103, Anaheim, California
  - Site Reference ID/Investigator# 16124, Los Angeles, California
  - Site Reference ID/Investigator# 16102, Orlando, Florida
  - Site Reference ID/Investigator# 16105, Baton Rouge, Louisiana
  - Site Reference ID/Investigator# 16106, Chapel Hill, North Carolina
  - Site Reference ID/Investigator# 16107, Dallas, Texas
  - Site Reference ID/Investigator# 16123, San Antonio, Texas
- Site Reference ID/Investigator# 16182, Santurce, Puerto Rico

REFERENCES:
- [Background] Mensing S, Polepally AR, Konig D, Khatri A, Liu W, Podsadecki TJ, Awni WM, Menon RM, Dutta S. Population Pharmacokinetics of Paritaprevir, Ombitasvir, Dasabuvir, Ritonavir, and Ribavirin in Patients with Hepatitis C Virus Genotype 1 Infection: Combined Analysis from 9 Phase 1b/2 Studies. AAPS J. 2016 Jan;18(1):270-80. doi: 10.1208/s12248-015-9846-1. Epub 2015 Nov 23. PMID 26597291
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Started | 8 | 8 | 8 | 6
Completed | 8 | 7 | 8 | 5
Not Completed | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were summarized by treatment group for all participants who received at least 1 dose of study drug. The treatment groups were compared with 1-way analysis of variance (ANOVA).
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV | Total
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (9.62) | 44.6 (12.96) | 47.8 (9.50) | 48.2 (7.31) | 46.5 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 1 | 9
  Male | 7 | 5 | 4 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximal Change From Baseline in Hepatitis C Virus Ribonucleic Acid (HCV RNA) Levels During ABT-333 Monotherapy Treatment
Description: Serum hepatitis C virus ribonucleic acid (HCV RNA) levels (reported as log10 IU/mL) were determined for each sample using a real-time reverse transcriptase polymerase chain reaction (RT-PCR) assay. The baseline value was the HCV RNA measurement before the first dose of ABT-333 on Day 1. The maximal change during monotherapy was nadir minus the baseline log10 HCV RNA level. Nadir was defined as the lowest log10 HCV RNA level any time after the first dose of study drug on Day 1 through the last log10 HCV RNA level before the first dose of study drug on Day 3. Data are reported as the least squares mean change from nadir ± standard error.
Time Frame: Prior to the first dose on Day 1 to before first dose on Day 3
Population: Participants received at least 1 dose of study drug and had at least 1 post-baseline measurement of HCV RNA.
Measure: Least Squares Mean (Standard Error); unit: log10 IU/mL
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 6
log10 IU/mL | -1.01 (0.18) | -0.78 (0.18) | -0.68 (0.18) | -0.26 (0.21)
Statistical Analysis 1: Comparison: ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Eight participants per ABT-333 group and 12 participants in the placebo group provided >95% power to detect a 1.4 log10 difference with a common standard deviation of 0.7 log10 using a two-sided, non-paired t-test with a significance level of 0.05; Test type: Superiority or Other; p = 0.012, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate
Statistical Analysis 2: Comparison: ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.071, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate
Statistical Analysis 3: Comparison: ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.140, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate

2. Primary Outcome: Mean Maximal Change From Baseline in Hepatitis C Virus Ribonucleic Acid (HCV RNA) Levels Through Day 28
Description: Serum hepatitis C virus ribonucleic acid (HCV RNA) levels (reported as log10 IU/mL) were determined for each sample using a real-time reverse transcriptase polymerase chain reaction (RT-PCR) assay. The baseline value was the HCV RNA measurement before the first dose of ABT-333 on Day 1. The maximal change during treatment was nadir minus the baseline log10 HCV RNA level. Nadir was defined as the lowest log10 HCV RNA level any time after the first dose of study drug on Day 1 through the last log10 HCV RNA level on Day 28. Data are reported as the least squares mean change from nadir ± standard error.
Time Frame: Prior to the first dose on Day 1 through Day 28
Population: Participants received at least 1 dose of study drug and had at least 1 post-baseline measurement of HCV RNA.
Measure: Least Squares Mean (Standard Error); unit: log10 IU/mL
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 6
log10 IU/mL | -3.65 (0.51) | -3.96 (0.51) | -3.59 (0.51) | -1.37 (0.59)
Statistical Analysis 1: Comparison: ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.008, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate
Statistical Analysis 2: Comparison: ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate
Statistical Analysis 3: Comparison: ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.009, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of ABT-333
Description: Blood samples were collected pre-dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and pre-dose on Day 2. The samples were analyzed for the concentration of ABT-333 using validated analytical methods. The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that a drug achieves in the blood after administration in a dosing interval. The Cmax of ABT-333 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: Pre-dose (time 0 hours); 2, 4, 8, 12, and 16 hours post-dose on Day 1; and pre-dose on Day 2
Population: Participants received at least 1 dose of study drug and had sufficient concentrations to characterize the pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 883 (575) | 1236 (724) | 1975 (619)

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of ABT-333
Description: Blood samples were collected pre-dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and pre-dose on Day 2. The samples were analyzed for the concentration of ABT-333 using validated analytical methods. The time to maximum plasma concentration (Tmax; measured in hours) is the time it takes for a drug to achieve Cmax. The Tmax of ABT-333 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: Pre-dose (time 0 hours); 2, 4, 8, 12, and 16 hours post-dose on Day 1; and pre-dose on Day 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
Hours | 3.80 (0.71) | 3.50 (0.93) | 3.50 (0.93)

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 12 Hours Post-dose (AUC12) of ABT-333
Description: Blood samples were collected pre-dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and pre-dose on Day 2. The samples were analyzed for the concentration of ABT-333 using validated analytical methods. The area under the plasma concentration-time curve (AUC; measured in ng*hr/mL) measures the total exposure of a drug in blood plasma. The AUC12 of ABT-333 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: Pre-dose (time 0 hours); 2, 4, 8, 12, and 16 hours post-dose on Day 1; and pre-dose on Day 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL | 5852 (4159) | 7548 (4016) | 12411 (4122)

6. Primary Outcome: Serum Concentrations of Pegylated Interferon (pegIFN)
Description: Blood samples were collected prior to the morning dose on Day 3; 4 hours after the morning dose on Day 3; prior to the morning dose on Days 4 and 5; and single samples were collected on Days 10, 17, 24, and 28. The samples were analyzed for the concentration of pegIFN (measured in ng/mL) using validated analytical methods and estimated using non-compartmental methods. Data are reported as the mean ± standard deviation.
Time Frame: Prior to the morning dose on Day 3; 4 hours after the morning dose on Day 3; prior to the morning dose on Days 4 and 5; and single samples were collected on Days 10, 17, 24, and 28
Population: Participants received at least 1 dose of study drug and had sufficient concentrations to characterize the pharmacokinetic parameters. When a different number of participants at a specific timepoint was used to analyze the data in the outcome measure, the n (number of participants) for each arm is denoted in the Category Title.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 6
ng/mL
  Prior to morning dose on Day 3 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  4 hours after morning dose on Day 3 (n=7, 8, 8, 6) | 0.70 (0.67) | 1.36 (1.51) | 0.09 (0.25) | 0.58 (0.70)
  Day 4 (n=8, 8, 7, 6) | 6.96 (4.04) | 6.51 (5.15) | 4.95 (4.50) | 3.42 (2.11)
  Day 5 | 9.06 (5.15) | 7.91 (4.82) | 5.57 (4.29) | 4.85 (3.17)
  Day 10 | 7.91 (2.21) | 6.47 (3.18) | 4.72 (3.28) | 4.48 (2.77)
  Day 17 (n=8, 8, 8, 5) | 12.3 (3.99) | 9.26 (4.28) | 8.73 (5.92) | 7.05 (5.06)
  Day 24 (n=8, 7, 8, 5) | 12.8 (3.45) | 12.1 (4.78) | 12.1 (7.11) | 8.58 (6.45)
  Day 28 (n=8, 7, 8, 5) | 17.4 (4.67) | 17.3 (3.95) | 17.0 (10.1) | 14.3 (10.0)

7. Primary Outcome: Plasma Concentrations of Ribavirin (RBV)
Description: Blood samples were collected prior to the morning dose on Day 3; 4 hours after the morning dose on Day 3; prior to the morning dose on Days 4 and 5; and single samples were collected on Days 10, 17, 24, and 28. The samples were analyzed for the concentration of RBV (measured in ng/mL) using validated analytical methods and estimated using non-compartmental methods. Data are reported as the mean ± standard deviation.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 6
ng/mL
  Prior to morning dose on Day 3 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  4 hours after morning dose on Day 3 | 0.46 (0.16) | 0.61 (0.40) | 0.51 (0.15) | 0.54 (0.19)
  Day 4 (n=5, 7, 5, 5) | 0.33 (0.07) | 0.46 (0.11) | 0.29 (0.17) | 0.36 (0.05)
  Day 5 (n=6, 6, 8, 5) | 0.61 (0.10) | 0.69 (0.22) | 0.48 (0.20) | 0.55 (0.14)
  Day 10 (n=7, 8, 8, 6) | 1.05 (0.17) | 1.24 (0.29) | 1.02 (0.38) | 1.05 (0.21)
  Day 17 (n=8, 8, 8, 5) | 1.47 (0.29) | 1.67 (0.40) | 1.32 (0.36) | 1.34 (0.52)
  Day 24 (n=8, 7, 8, 5) | 1.76 (0.31) | 1.91 (0.38) | 1.60 (0.39) | 1.49 (0.19)
  Day 28 (n=8, 7, 8, 5) | 1.76 (0.44) | 2.07 (0.53) | 1.56 (0.46) | 1.68 (0.66)

8. Primary Outcome: Number of Participants Having Treatment-emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence that did not have a causal relationship with treatment. An Adverse Drug Reaction (ADR) was any noxious and undesired reaction related to the experimental drug or experiment. A serious adverse event (SAE) was an AE that resulted in death, was life-threatening, resulted in or prolonged hospitalization, resulted in congenital anomaly, was persistent or caused significant disability/incapacity, spontaneous or elective abortion, or required intervention to prevent a serious outcome. AEs were rated for severity as either:
  1. Mild - transient and easily tolerated;
  2. Moderate - caused discomfort and interrupted usual activities;
  3. Severe - caused considerable interference with usual activities, may be incapacitating or life-threatening.
  AEs related to direct-acting antiviral agents (DAAs) were assessed as being either probably or possibly related by the investigator.
Time Frame: AEs were collected from the time of study drug administration to 30 days after last dose of study drug (8 Weeks)
Population: Participants received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 6
participants
  Any AE | 8 | 8 | 8 | 5
  Any AE at least possibly drug related | 4 | 3 | 2 | 1
  Any severe AE | 1 | 0 | 0 | 0
  Any serious AE | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of study drug | 0 | 0 | 0 | 0
  Any fatal events | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Hepatitis C Virus Ribonucleic Acid (HCV RNA) Levels Through Day 28 or Final Visit
Description: Serum hepatitis C virus ribonucleic acid (HCV RNA) levels (reported as log10 IU/mL) were determined using a real-time reverse transcriptase polymerase chain reaction (RT-PCR) assay. The baseline value was the HCV RNA measurement before the first dose of ABT-333 on Day 1 and the Day 28 or Final Visit value was the last HCV RNA measurement during the study. Data are reported as the least squares mean change from baseline ± standard error.
Time Frame: Day 28 and Final Visit
Population: Participants received at least 1 dose of study drug and had at least 1 post-baseline measurement of HCV RNA. When a different number of participants at a specific timepoint was used to analyze the data in the outcome measure, the n (number of participants) for each arm is denoted in the Category Title.
Measure: Least Squares Mean (Standard Error); unit: log10 IU/mL
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 6
log10 IU/mL
  Day 28 (n=8, 7, 7, 5) | -3.65 (0.53) | -3.67 (0.57) | -3.24 (0.57) | -1.45 (0.68)
  Final Visit | -3.65 (0.53) | -3.86 (0.53) | -3.48 (0.53) | -1.35 (0.61)
Statistical Analysis 1: Comparison: ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; The statistical analysis represents the Day 28 time point; Test type: Superiority or Other; p = 0.018, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate
Statistical Analysis 2: Comparison: ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; The statistical analysis represents the Day 28 time point; Test type: Superiority or Other; p = 0.020, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate
Statistical Analysis 3: Comparison: ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; The statistical analysis represents the Day 28 time point; Test type: Superiority or Other; p = 0.054, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate
Statistical Analysis 4: Comparison: ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; The statistical analysis represents the Final Visit time point; Test type: Superiority or Other; p = 0.010, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate
Statistical Analysis 5: Comparison: ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; The statistical analysis represents the Final Visit time point; Test type: Superiority or Other; p = 0.005, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate
Statistical Analysis 6: Comparison: ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; The statistical analysis represents the Final Visit time point; Test type: Superiority or Other; p = 0.014, ANCOVA — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05; The treatment group was the factor and log10 baseline HCV RNA level was the covariate

10. Secondary Outcome: Percentage of Participants With at Least a 2 log10 Maximal Decrease in Hepatitis C Virus Ribonucleic Acid (HCV RNA) Levels During ABT-333 Treatment
Description: Serum hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined using a real-time reverse transcriptase polymerase chain reaction (RT-PCR) assay. The baseline value was the HCV RNA measurement before the first dose of ABT-333 on Day 1. Data are reported as the percentage of participants.
Time Frame: Prior to the first dose on Day 1 and Day 28
Population: Participants received at least 1 dose of study drug and had at least 1 post-baseline measurement of HCV RNA.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 6
percentage of participants | 87.5 | 87.5 | 62.5 | 16.7
Statistical Analysis 1: Comparison: ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.026, Fisher Exact — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05
Statistical Analysis 2: Comparison: ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.026, Fisher Exact — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05
Statistical Analysis 3: Comparison: ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.138, Fisher Exact — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05

11. Secondary Outcome: Percentage of Participants With Hepatitis C Virus Ribonucleic Acid (HCV RNA) Levels ≤ 25 IU/mL (the Lower Limit of Quantitation [LLOQ]) at Day 28 or Final Visit
Description: Serum hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined for each sample using a real-time reverse transcriptase polymerase chain reaction (RT-PCR) assay. The lower limit of quantification (LLOQ) was defined as HCV RNA levels ≤ 25 IU/mL. Data are reported as the percentage of participants.
Time Frame: Day 28 or Final Visit
Population: Participants received at least 1 dose of study drug and had at least 1 post-baseline measurement of hepatitis C virus ribonucleic acid (HCV RNA).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 6
percentage of participants | 37.5 | 25.0 | 62.5 | 0.00
Statistical Analysis 1: Comparison: ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.209, Fisher Exact — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05
Statistical Analysis 2: Comparison: ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.473, Fisher Exact — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05
Statistical Analysis 3: Comparison: ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.031, Fisher Exact — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05

12. Secondary Outcome: Percentage of Participants With Hepatitis C Virus Ribonucleic Acid (HCV RNA) Levels ≤ 10 IU/mL (Lower Limit of Detection [LLOD]) at Day 28 or Final Visit
Description: Serum hepatitis C virus ribonucleic acid (HCV RNA) levels (measured in IU/mL) were determined for each sample using a real-time reverse transcriptase polymerase chain reaction (RT-PCR) assay. The lower limit of detection (LLOD) was defined as a HCV RNA level equal to 10 IU/mL. Data are reported as the percentage of participants.
Time Frame: Day 28 or Final Visit
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 6
percentage of participants | 37.5 | 0.00 | 12.5 | 0.00
Statistical Analysis 1: Comparison: ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.209, Fisher Exact — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05
Statistical Analysis 2: Comparison: ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 1.000, Fisher Exact — No adjustments were made for multiple comparisons and the pre-specified, two-sided significance level was 0.05

13. Secondary Outcome: Number of Participants With Resistance-Associated Variants in Non-structural Viral Protein 5B (NS5B) Through Day 28
Description: Samples from Days 1, 5, 10, 17, 24 and 28 were analyzed for the presence of resistance-associated amino acids using population sequencing and compared to the baseline non-structural viral protein 5B (NS5B) sequence to assess amino acid changes. The amino acid sequence of NS5B before the first dose of ABT-333 on Day 1 was defined as the baseline sequence. The number of participants with variants at resistance-associated amino acid positions in the post-baseline samples are presented.
Time Frame: Days 1, 5, 10, 17, 24 and 28
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
participants
  Day 1 | 0 | 1 | 0
  Day 5 (n=6, 8, 7) | 1 | 1 | 1
  Day 10 (n=6, 6, 7) | 1 | 1 | 2
  Day 17 (n=5, 5, 6) | 2 | 2 | 2
  Day 24 (n=3, 3, 2) | 3 | 3 | 1
  Day 28 (n=4, 3, 3) | 2 | 2 | 3

14. Secondary Outcome: Number of Participants With Maximal Phenotypic Resistance to ABT-333 >10 Fold Relative to Baseline Through Day 28
Description: Phenotypic resistance to ABT-333 was assessed by calculating the fold difference in the half maximal effective concentration (EC50) compared with the EC50 for the corresponding baseline sample, and the maximal fold change in EC50 from baseline over the Day 5-28 period. The resistance sample drawn before the first dose of ABT-333 on Day 1 was defined as the baseline sample. The number of participants with phenotypic resistance in the post-baseline samples are presented.
Time Frame: Days 1 through 28
Population: Participants received at least 1 dose of study drug and had at least 1 post-baseline measurement of HCV RNA.
Measure: Number; unit: participants
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (600 mg) Twice Daily (BID) + pegIFN/RBV | ABT-333 (1200 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
participants | 4 | 4 | 5

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of study drug administration to 30 days after last dose of study drug ( 8 Weeks); SAEs were also collected from the time that informed consent was obtained to 30 days after last dose of study drug (up to 12 weeks).
Groups:
- ABT-333 (300 mg) Twice Daily (BID) + (pegIFN/RBV): Hepatitis C virus (HCV) positive, treatment-naive participants received 300 mg ABT-333 BID for 2 days followed by 300 mg ABT-333 BID with pegylated interferon/ribavirin (pegIFN/RBV) for 26 days. Pegylated interferon was administered at 180 μg subcutaneously once a week and the RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-333 (600 mg) Twice Daily (BID) + (pegIFN/RBV): Hepatitis C virus (HCV) positive, treatment-naive participants received 600 mg ABT-333 BID for 2 days followed by 600 mg ABT-333 BID with pegylated interferon/ribavirin (pegIFN/RBV) for 26 days. Pegylated interferon was administered at 180 μg subcutaneously once a week and the RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-333 (1200 mg) Once Daily (QD) + (pegIFN/RBV): Hepatitis C virus (HCV) positive, treatment-naive participants received 1200 mg ABT-333 QD for 2 days followed by 1200 mg ABT-333 BID with pegylated interferon/ribavirin (pegIFN/RBV) for 26 days. Pegylated interferon was administered at 180 μg subcutaneously once a week and the RBV was dosed 1000 or 1200 mg daily divided twice a day.
- Placebo + (pegIFN/RBV): Hepatitis C virus (HCV) positive, treatment-naïve participants received matching placebo once daily (QD) or twice daily (BID) for 2 days followed by placebo QD or BID with pegylated interferon/ribavirin (pegIFN/RBV) for 26 days. Pegylated interferon was administered at 180 μg subcutaneously once a week and the RBV was dosed 1000 or 1200 mg daily divided twice a day.
Arm/Group | ABT-333 (300 mg) Twice Daily (BID) + (pegIFN/RBV) | ABT-333 (600 mg) Twice Daily (BID) + (pegIFN/RBV) | ABT-333 (1200 mg) Once Daily (QD) + (pegIFN/RBV) | Placebo + (pegIFN/RBV)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-333 (300 mg) Twice Daily (BID) + (pegIFN/RBV) (N=8) | ABT-333 (600 mg) Twice Daily (BID) + (pegIFN/RBV) (N=8) | ABT-333 (1200 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | Placebo + (pegIFN/RBV) (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 3 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 1
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 | 0 | 0 | 1
EYE PRURITUS (Eye disorders) | 1 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 1 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 1 | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GLOSSODYNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 2 | 3 | 0
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1 | 1 | 0
CHILLS (General disorders) | 2 | 1 | 1 | 0
FATIGUE (General disorders) | 5 | 1 | 1 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 2 | 3 | 3
IRRITABILITY (General disorders) | 1 | 1 | 0 | 2
MALAISE (General disorders) | 1 | 0 | 0 | 0
PAIN (General disorders) | 0 | 0 | 1 | 0
PYREXIA (General disorders) | 2 | 0 | 2 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
JOINT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
ANOREXIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 1 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 5 | 5 | 4 | 2
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 2 | 1
INSOMNIA (Psychiatric disorders) | 1 | 1 | 0 | 1
MOOD SWINGS (Psychiatric disorders) | 0 | 0 | 1 | 0
POLYURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.